CLINICAL TRIAL: NCT07304765
Title: The Acute Effects of Neurodynamic Stretching the Shear Wave Velocity: on Application on Muscle and Nerve Tissues
Brief Title: Acute Effects of Neurodynamic Stretching on Muscle-tendon Complex
Acronym: ELASTRETCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, Nicolas Babault, Prof, University of Burgundy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CEP2204
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Stretching; Control Condition
Keywords: stretching; stiffness; nerve; muscle; flexibility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control (No Intervention): Seated at rest during the same duration than the interventions
- Static stretching at pain threshold (Active Comparator): Static stretching at pain threshold of the right hamstring muscles 5x60s with 20s rest
  Interventions: Other: Maximal static stretching
- Neurodynamic tensioning at pain threshold (Experimental): Neurodynamic tensioning of the right hamstring muscles 5x60s with 20s rest at pain threshold
  Interventions: Other: Maximal neurodynamic tensioning
- Neurodynamic flossing at pain threshold (Experimental): Neurodynamic flossing of the right hamstring muscles 5x60s with 20s rest at pain threshold
  Interventions: Other: Maximal neurodynamic flossing
- Static stretching at submaximal intensity (Active Comparator): Static stretching of the right hamstring muscles 5x60s with 20s rest at 10% below pain threshold
  Interventions: Other: Submaximal static stretching
- Neurodynamic tensioning at submaximal intensity (Active Comparator): Neurodynamic tensioning stretching of the right hamstring muscles 5x60s with 20s rest at 10% below pain threshold
  Interventions: Other: Submaximal neurodynamic tensioning
- Neurodynamic flossing at submaximal intensity (Active Comparator): Neurodynamic flossing stretching of the right hamstring muscles 5x60s with 20s rest at 10% below pain threshold
  Interventions: Other: Submaximal neurodynamic flossing

INTERVENTIONS:
Other: Maximal static stretching — Static stretching was applied at pain threshold on hamstring muscles and repeated 5 times during 60s at the point of pain. Static stretching mainly focused muscle-tendon tissues.
  Arms: Static stretching at pain threshold
Other: Submaximal static stretching — Static stretching was applied 10% below pain threshold on hamstring muscles and repeated 5 times during 60s at the point of pain. Static stretching mainly focused muscle-tendon tissues.
  Arms: Static stretching at submaximal intensity
Other: Maximal neurodynamic tensioning — Neurodynamic tensioning was applied at pain threshold on hamstring muscles and repeated 5 times during 60s at the point of pain. During the neurodynamic conditions, head and ankle movement permitted to mobilize nerve tissues. Tensioning is maintaining the position.
  Arms: Neurodynamic tensioning at pain threshold
Other: Submaximal neurodynamic tensioning — Neurodynamic tensioning was applied 10% below pain threshold on hamstring muscles and repeated 5 times during 60s at the point of pain. During the neurodynamic conditions, head and ankle movement permitted to mobilize nerve tissues. Tensioning is maintaining the position.
  Arms: Neurodynamic tensioning at submaximal intensity
Other: Maximal neurodynamic flossing — Neurodynamic flossing was applied at pain threshold on hamstring muscles and repeated 5 times during 60s at the point of pain. During the neurodynamic conditions, head and ankle movement permitted to mobilize nerve tissues. Flossing is the alternation of these movements every 2 seconds.
  Arms: Neurodynamic flossing at pain threshold
Other: Submaximal neurodynamic flossing — Neurodynamic flossing was applied 10% below pain threshold on hamstring muscles and repeated 5 times during 60s at the point of pain. During the neurodynamic conditions, head and ankle movement permitted to mobilize nerve tissues. Flossing is the alternation of these movements every 2 seconds.
  Arms: Neurodynamic flossing at submaximal intensity

SUMMARY:
Neurodynamic mobilization techniques are widely applied in rehabilitation and physiotherapy to enhance the mobility and function of peripheral nerves. Two main approaches are distinguished. Nerve tensioning and nerve flossing. They both involve proximal and distal joint movements to induce greater neural sliding while avoiding excessive tensile stress. However, contradictory findings on neurodynamic techniques highlighted the current lack of consensus regarding these techniques. Moreover, neurodynamic techniques are of interest for patients, it appeared it could also be applied in healthy individuals and more particularly in athletes. Accordingly, the primary objective of the present study was to determine the immediate effect of two neurodynamic mobilization techniques (flossing vs. tensioning) on the sciatic nerve and hamstring tissues using the shear wave elastography (SWE, a form of ultrasonography).

DETAILED DESCRIPTION:
Neurodynamic mobilization techniques are frequently applied in rehabilitation settings to enhance the mobility and function of peripheral nerves, particularly in the management of neuropathic pain such as carpal tunnel syndrome, radiculopathies, or sciatica. Two main approaches are distinguished. Nerve tensioning involves maintaining the nerve stretched at the end of the joint range of motion with relatively limited excursion. It is similar to a static stretching intervention but with distal (ankle) and proximal (cervical) tensions. Nerve flossing (also termed gliding or sliders), consists of alternating proximal and distal joint movements to induce greater neural sliding while avoiding excessive tensile stress. However, contradictory findings on neurodynamic techniques highlighted the current lack of consensus regarding the acute effects of the different possible neurodynamic techniques on sciatic nerves, particularly in healthy tissues. Moreover, neurodynamic techniques are of interest for patients, it appeared it could also be applied in healthy individuals and more particularly in athletes. Performed in patients, healthy or athletes, no study has compared both tensioning or flossing techniques. Moreover, because these techniques involved nerve mobilisation, the intensity should have a main effect of its efficiency. Accordingly, the primary objective of the present study was to determine the immediate effect of two neurodynamic mobilization techniques (flossing vs. tensioning) on the sciatic nerve and hamstring tissues using the shear wave elastography (SWE). This method has been shown reliable to provide non-invasive real-time assessments of soft tissues elastic properties. The secondary aim was to determine the effects of stretching intensity (at the point of pain threshold or below).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* physical active
* no injuries (lower limb or back pain) in the past 3 months

Exclusion Criteria:

* Specific lower limb (hamstring) injuries in the past 2 years
* Not restraining activity 24h before participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Nerve shear wave velocity using elastography | Before the intervention and at the end (immediately after) the intervention
  Shear wave velocity of the sciatic nerve will be evaluated by using an ultrasound (echography) device with a specific mode called "shear wave elastography". Briefly, the ultrasound probe will deliver an ultrasound wave. The propagation speed (called '"shear wave velocity") will be measured by the same probe. The greater the velocity is, the harder the tissue is.

SECONDARY OUTCOMES:
Muscle shear wave velocity using elastography | Before the intervention and at the end (immediately after) the intervention
  Shear wave velocity of the biceps femoris muscle will be evaluated by using an ultrasound (echography) device with a specific mode called "shear wave elastography". Briefly, the ultrasound probe will deliver an ultrasound wave. The propagation speed (called '"shear wave velocity") will be measured by the same probe. The greater the velocity is, the harder the tissue is.
Hamstring force | Before the intervention and at the end (immediately after) the intervention
  Maximal torque during a maximal voluntary hamstring contraction
Biceps femoris activity | Before the intervention and at the end (immediately after) the intervention
  Electromyographic activity of biceps femoris muscle
Semitendinosus activity | Before the intervention and at the end (immediately after) the intervention
  Electromyographic activity of semitendinosus
passive knee extension | Before the intervention and at the end (immediately after) the intervention
  The final passive range of motion of the hamstring muscles
Global flexibility | Before the intervention and at the end (immediately after) the intervention
  the stand and reach test to evaluate flexibility (in centimeters)
Slump test | Before the intervention and at the end (immediately after) the intervention
  Seated flexibility using the slump test (in degrees)
discomfort | At the end (immediately after) the intervention
  rating of perceived discomfort during the intervention (from 1 to 10, no discomfort to maximal discomfort, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Babault, PhD, Principal Investigator — Universite Bourgogne Europe - Sport Science Faculty
Locations (1):
- Universite Bourgogne Europe - faculty of sports sciences, Dijon, France

IPD SHARING:
Plan to Share IPD: Yes
data freely available in online websites